CLINICAL TRIAL: NCT02034877
Title: A Phase 4/3, Open-label, Single-arm, Multicenter Study To Describe The Safety And Immunogenicity Of 13-valent Pneumococcal Conjugate Vaccine In Adults 50 To 65 Years Of Age And In Children 6 To 17 Years Of Age In India
Brief Title: 13-valent Pneumococcal Conjugate Vaccine Study in Adults and Children in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: B1851140; 2014-001174-34 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Prevention of Pneumonia and Invasive Disease Caused by the Serotypes in 13vPnC
Keywords: 13-valent pneunococcal conjugate vaccine; pneumococcal disease prevention; safety and immunogenicity study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal conjugate vaccine; Procedure: Blood sample collection

INTERVENTIONS:
Biological: 13-valent Pneumococcal conjugate vaccine — 1 dose (0.5 mL/ pre-filed syringe) of 13vPnC administered at visit 1
Procedure: Blood sample collection — 10 mL of blood will be collected just before and approximately 1 month after vaccination.

SUMMARY:
This study is to describe the safety and immunogenicity of 13vPnC in Indian adults 50 to 65 years of age and in Indian children 6 to 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

Indian adults subjects between 50 and 65 years of age and indian children between 6 and 17years of age, determined by clinical judgment to be eligible for 13vPnC vaccination.

Exclusion Criteria:

Any contraindication to 13vPnC vaccination, vaccination with any pneumococcal vaccine within the last year

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- India (16):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - B. J. Medical College & Civil Hospital, Ahmedabad, Gujarat
  - S.B.K.S Medical Institute & Research Centre, Vadodara, Gujarat
  - M.S. Ramaiah Cliical Research Centre, M.S. Ramaiah Medical College & Hospitals, Bangalore, Karnataka
  - M.S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Sushruta Multispeciality Hospital & Research Centre Pvt. Ltd., Hubli, Karnataka
  - Cheluvamba Hospital, Mysore, Karnataka
  - Niramaya Hospital, Chinchwad Pune, Maharashtra
  - Supe Heart & Diabetes Hospital and Research Centre, Nashik, Maharashtra
  - Chopda Medicare and Research Centre Pvt. Ltd, Nashik, Maharashtra
  - Medipoint Hospitals Pvt. Ltd., Pune, Maharashtra
  - Padmashree Dr. D. Y. Patil Medical College, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
  - Samvedna Hospital, Varanasi, Uttar Pradesh
  - Bhatia Hospital, Mumbai
  - Orange City Hospital and Research Institute, Nagpur

REFERENCES:
- [Derived] Solanki BB, Juergens C, Chopada MB, Supe P, Sundaraiyer V, Le Dren-Narayanin N, Cutler MW, Gruber WC, Scott DA, Schmoele-Thoma B. Safety and immunogenicity of a 13-valent pneumococcal conjugate vaccine in adults 50 to 65 years of age in India: An open-label trial. Hum Vaccin Immunother. 2017 Sep 2;13(9):2065-2071. doi: 10.1080/21645515.2017.1331796. PMID 28881165
- [Derived] Agarkhedkar S, Juergens C, Balasundaram K, Agarkhedkar S, Sundaraiyer V, Le Dren-Narayanin N, Cutler MW, Gruber WC, Scott DA, Schmoele-Thoma B; B1851140 Study Team. Safety and Immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine in Children 6-17 Years of Age in India: An Open-label Trial. Pediatr Infect Dis J. 2017 Nov;36(11):e283-e285. doi: 10.1097/INF.0000000000001695. PMID 28719496
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851140&StudyName=13-valent%20pneumococcal%20conjugate%20vaccine%20study%20in%20adults%20and%20children%20in%20India%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1200 (200 pediatric and 1000 adult) participants were randomized in the study. Out of the 1000 adult participants, 999 participants and all 200 pediatric participants received vaccination.
Groups:
- 13vPnC (Pediatric Participants): Pediatric participants aged 6 to 17 years received 1 single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly.
- 13vPnC (Adult Participants): Adult participants aged 50 to 65 years received 1 single 0.5 mL dose of 13vPnC intramuscularly.
Period: Overall Study
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Started | 200 | 999
Completed | 200 | 993
Not Completed | 0 | 6
Not completed — Lost to Follow-up | 0 | 3
Not completed — No Longer Willing to Participate | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received 1 dose of 13vPnC vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants) | Total
Number analyzed (Participants) | 200 | 999 | 1199
Age, Customized [Number; unit: Participants]
  6 to 11 years | 157 | 0 | 157
  12 to 17 years | 43 | 0 | 43
  50 to 64 years | 0 | 997 | 997
  65 to 84 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 414 | 521
  Male | 93 | 585 | 678

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) Within 1 Month After 13vPnC Vaccination
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 1 month after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Within 1 month after 13vPnC vaccination
Population: Safety population included all participants who received 1 dose of 13vPnC vaccination.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 999
Percentage of participants
  AEs | 0 | 7
  SAEs | 0 | 0

2. Primary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) Before 13vPnC Vaccination
Description: Antibody-mediated opsonophagocytic activity against each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were measured using a quantitative functional OPA assay. OPA titers were expressed as the reciprocal of the highest serum dilution that reduces survival of the pneumococci by at least 50 percent (%). For each serotype, GMTs were calculated using the logarithmically transformed assay results. Confidence intervals (CIs) for GMTs were back transformations of a CI based on the Student t distribution for the mean of the logarithmically transformed assay results. Here, number of participants analyzed (N) signifies participants evaluable for this outcome measure.
Time Frame: Before 13vPnC vaccination
Population: Evaluable immunogenicity population: eligible participants received 13vPnC;had blood drawn within pre-specified time-frames with at least 1 valid,determinate assay result,no major protocol violation. Only 400 adults were selected for immunogenicity analysis, 'n'=number of participants with valid and determinate assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 388
Titers
  Serotype 1 (n=194, 385) | 11 [9.6 to 11.8] | 11 [10.4 to 11.7]
  Serotype 3 (n=197, 384) | 18 [15.3 to 22.2] | 10 [9.1 to 11.1]
  Serotype 4 (n=176, 358) | 230 [155.8 to 339.2] | 212 [165.7 to 271.3]
  Serotype 5 (n=199, 383) | 19 [16.8 to 20.9] | 17 [16.5 to 18.3]
  Serotype 6A (n=170, 347) | 461 [339.6 to 626.8] | 304 [255.0 to 363.5]
  Serotype 6B (n=163, 339) | 263 [184.2 to 376.3] | 331 [266.2 to 410.4]
  Serotype 7F (n=160, 363) | 742 [585.8 to 940.5] | 324 [289.0 to 363.9]
  Serotype 9V (n=183, 369) | 2097 [1702.4 to 2582.9] | 826 [730.8 to 933.4]
  Serotype 14 (n=182, 380) | 1387 [1091.0 to 1763.0] | 400 [335.9 to 476.3]
  Serotype 18C (n=154, 374) | 216 [138.9 to 336.6] | 213 [170.7 to 265.8]
  Serotype 19A (n=195, 383) | 62 [47.2 to 80.1] | 66 [56.4 to 76.2]
  Serotype 19F (n=194, 375) | 265 [201.9 to 348.5] | 115 [97.2 to 136.2]
  Serotype 23F (n=184, 379) | 84 [58.3 to 121.4] | 57 [45.5 to 71.3]

3. Primary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After 13vPnC Vaccination
Description: Antibody-mediated opsonophagocytic activity against each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were measured using a quantitative functional OPA assay. OPA titers were expressed as the reciprocal of the highest serum dilution that reduces survival of the pneumococci by at least 50%. For each serotype, GMTs were calculated using the logarithmically transformed assay results. CIs for GMTs were back transformations of a CI based on the Student t distribution for the mean of the logarithmically transformed assay results. Here, number of participants analyzed (N) signifies participants evaluable for this outcome measure.
Time Frame: 1 month after 13vPnC vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 388
Titers
  Serotype 1 (n=191, 376) | 176 [146.1 to 212.7] | 266 [231.4 to 304.6]
  Serotype 3 (n=200, 378) | 118 [103.7 to 133.6] | 143 [126.4 to 162.4]
  Serotype 4 (n=199, 371) | 7860 [7074.0 to 8732.4] | 6029 [5433.0 to 6691.4]
  Serotype 5 (n=200, 354) | 286 [232.9 to 351.9] | 639 [540.5 to 755.4]
  Serotype 6A (n=199, 376) | 9247 [8197.4 to 10431.8] | 6653 [5963.1 to 7423.8]
  Serotype 6B (n=195, 362) | 6755 [6018.5 to 7581.7] | 7690 [6844.8 to 8640.2]
  Serotype 7F (n=199, 378) | 5251 [4787.9 to 5758.1] | 3211 [2939.4 to 3507.2]
  Serotype 9V (n=197, 375) | 7028 [6211.9 to 7951.1] | 5441 [4954.6 to 5974.5]
  Serotype 14 (n=197, 379) | 7484 [6586.1 to 8503.6] | 3182 [2789.9 to 3628.6]
  Serotype 18C (n=198, 360) | 8641 [7729.0 to 9661.2] | 7670 [6818.0 to 8627.4]
  Serotype 19A (n=197, 380) | 1928 [1660.6 to 2238.5] | 2371 [2092.7 to 2686.6]
  Serotype 19F (n=200, 368) | 3551 [3099.1 to 4069.0] | 3340 [2937.7 to 3797.3]
  Serotype 23F (n=199, 378) | 4419 [3945.7 to 4949.2] | 5766 [5034.4 to 6604.2]

4. Primary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) From Before 13vPnC Vaccination to 1 Month After 13vPnC Vaccination
Description: GMFRs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before 13vPnC vaccination to 1 month after 13vPnC vaccination were computed using the logarithmically transformed assay results. CIs for GMFRs were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before and after vaccination blood draws. Here, number of participants analyzed (N) signifies participants evaluable for this outcome measure.
Time Frame: Before 13vPnC vaccination, 1 month after 13vPnC vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 388
Fold rise
  Serotype 1 (n=185, 373) | 16.3 [13.26 to 19.92] | 24.0 [20.79 to 27.64]
  Serotype 3 (n=197, 374) | 6.4 [5.23 to 7.80] | 14.4 [12.49 to 16.63]
  Serotype 4 (n=175, 344) | 32.6 [21.59 to 49.08] | 27.6 [21.15 to 35.89]
  Serotype 5 (n=199, 351) | 15.3 [12.15 to 19.26] | 36.9 [31.18 to 43.60]
  Serotype 6A (n=169, 339) | 19.1 [13.77 to 26.48] | 23.1 [18.93 to 28.12]
  Serotype 6B (n=160, 316) | 24.9 [17.19 to 35.94] | 24.2 [19.35 to 30.27]
  Serotype 7F (n=160, 354) | 7.1 [5.52 to 9.05] | 9.5 [8.30 to 10.96]
  Serotype 9V (n=180, 358) | 3.3 [2.65 to 4.10] | 6.6 [5.75 to 7.48]
  Serotype 14 (n=179, 372) | 5.5 [4.16 to 7.19] | 7.8 [6.33 to 9.70]
  Serotype 18C (n=153, 350) | 41.5 [26.82 to 64.25] | 36.6 [28.69 to 46.68]
  Serotype 19A (n=192, 375) | 31.2 [23.38 to 41.74] | 36.3 [30.21 to 43.60]
  Serotype 19F (n=194, 358) | 13.3 [9.87 to 17.99] | 29.2 [23.64 to 35.98]
  Serotype 23F (n=183, 371) | 53.3 [36.17 to 78.40] | 102.7 [81.10 to 130.10]

5. Primary Outcome: Percentage of Participants With Opsonophagocytic Activity (OPA) Titer Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) Before 13vPnC Vaccination
Description: Percentage of participants achieving serotype-specific pneumococcal OPA titer >=LLOQ, along with the corresponding 95% CIs for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) are presented. Exact 2-sided CIs for the observed proportion of participants were calculated using Clopper and Pearson method. LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43; Pn7F, 210 (for adult participants); Pn7F, 113 (for pediatric participants) Pn09V, 345 (for adult participants); Pn09V, 141 (for pediatric participants); Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; Pn23F, 13. Here, number of participants analyzed (N) signifies participants evaluable for this outcome measure.
Time Frame: Before 13vPnC vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 388
Percentage of participants
  Serotype 1 (n=194, 385) | 6.7 [3.6 to 11.2] | 12.7 [9.6 to 16.5]
  Serotype 3 (n=197, 384) | 50.8 [43.6 to 57.9] | 25.8 [21.5 to 30.5]
  Serotype 4 (n=176, 358) | 60.2 [52.6 to 67.5] | 65.6 [60.5 to 70.6]
  Serotype 5 (n=199, 383) | 12.1 [7.9 to 17.4] | 13.1 [9.8 to 16.8]
  Serotype 6A (n=170, 347) | 73.5 [66.2 to 80.0] | 77.8 [73.1 to 82.1]
  Serotype 6B (n=163, 339) | 55.8 [47.9 to 63.6] | 68.7 [63.5 to 73.6]
  Serotype 7F (n=160, 363) | 78.1 [70.9 to 84.3] | 57.9 [52.6 to 63.0]
  Serotype 9V (n=183, 369) | 90.2 [84.9 to 94.1] | 74.5 [69.8 to 78.9]
  Serotype 14 (n=182, 380) | 91.2 [86.1 to 94.9] | 82.1 [77.9 to 85.8]
  Serotype 18C (n=154, 374) | 50.0 [41.8 to 58.2] | 67.6 [62.6 to 72.4]
  Serotype 19A (n=195, 383) | 62.1 [54.8 to 68.9] | 74.2 [69.5 to 78.5]
  Serotype 19F (n=194, 375) | 66.5 [59.4 to 73.1] | 54.4 [49.2 to 59.5]
  Serotype 23F (n=184, 379) | 53.3 [45.8 to 60.6] | 54.6 [49.5 to 59.7]

6. Primary Outcome: Percentage of Participants With Opsonophagocytic Activity (OPA) Titer Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ) 1 Month After 13vPnC Vaccination
Description: as for outcome 5
Time Frame: 1 month after 13vPnC vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Number analyzed (Participants) | 200 | 388
Percentage of participants
  Serotype 1 (n=191, 376) | 92.7 [88.0 to 95.9] | 94.9 [92.2 to 96.9]
  Serotype 3 (n=200, 378) | 99.5 [97.2 to 100.0] | 95.8 [93.2 to 97.6]
  Serotype 4 (n=199, 371) | 100.0 [98.2 to 100.0] | 100.0 [99.0 to 100.0]
  Serotype 5 (n=200, 354) | 91.0 [86.1 to 94.6] | 93.8 [90.7 to 96.1]
  Serotype 6A (n=199, 376) | 100.0 [98.2 to 100.0] | 100.0 [99.0 to 100.0]
  Serotype 6B (n=195, 362) | 100.0 [98.1 to 100.0] | 99.7 [98.5 to 100.0]
  Serotype 7F (n=199, 378) | 100.0 [98.2 to 100.0] | 99.2 [97.7 to 99.8]
  Serotype 9V (n=197, 375) | 100.0 [98.1 to 100.0] | 99.7 [98.5 to 100.0]
  Serotype 14 (n=197, 379) | 100.0 [98.1 to 100.0] | 98.7 [96.9 to 99.6]
  Serotype 18C (n=198, 360) | 100.0 [98.2 to 100.0] | 99.4 [98.0 to 99.9]
  Serotype 19A (n=197, 380) | 99.0 [96.4 to 99.9] | 99.5 [98.1 to 99.9]
  Serotype 19F (n=200, 368) | 99.0 [96.4 to 99.9] | 98.9 [97.2 to 99.7]
  Serotype 23F (n=199, 378) | 100.0 [98.2 to 100.0] | 98.9 [97.3 to 99.7]

ADVERSE EVENTS:
Time Frame: Baseline to 1 month after 13vPnC vaccination (up to 42 days)
Arm/Group | 13vPnC (Pediatric Participants) | 13vPnC (Adult Participants)
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/999
Other Adverse Events (participants affected / at risk) | 0/200 | 70/999
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (Pediatric Participants) (N=200) | 13vPnC (Adult Participants) (N=999)
Nausea (Gastrointestinal disorders) | 0 | 1
Vaccination site pain (General disorders) | 0 | 46
Pyrexia (General disorders) | 0 | 22
Fatigue (General disorders) | 0 | 4
Chills (General disorders) | 0 | 2
Vaccination site erythema (General disorders) | 0 | 2
Vaccination site nodule (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Vaccination site induration (General disorders) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.